CLINICAL TRIAL: NCT06865586
Title: A Comparative Study of Tumor Specific Mesocolic Excision and Complete Mesocolic Excision for Right Sided Colon Cancer : Asian Multicenter Retrospective Study
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Korea University Anam Hospital (Other); Kyungpook National University Chilgok Hospital (Other); Severance Hospital (Other); Chinese University of Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); North District Hospital (Other); China Medical University Hospital (Other)
Responsible Party: Principal Investigator, In Ja Park, Professor, Asan Medical Center
Other Study IDs: SMART core
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer; Lymph Node Dissection; Laparoscopic Colon Surgery; Robotic Surgical Procedure
Keywords: colon cancer; right hemicolectomy; complete mesocolic excision; lymph node dissection; microinvasive surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent laparoscopic or robotic right hemicolectomy with CME from 2015 to 2020: Patients who underwent laparoscopic or robotic right hemicolectomy with Complete mesocolic excision from 2015 to 2020 in 8 centers
- Patients who underwent with tumor specific mesocolic exicision from 2015 to 2020: Patients who underwent laparoscopic or robotic right hemicolectomy with tumor specific mesocolic exicision from 2015 to 2020 in 8 centers

SUMMARY:
The goal of this observational study is to determine the optimal surgical strategy based on oncologic outcomes in patients with stage I-III right-sided colon cancer who underwent curative right hemicolectomy.

The main question it aims to answer is: Is there a significant difference in 5-year recurrence-free survival (RFS) between patients treated with Complete Mesocolic Excision (CME) and those treated with tumor specific mesocolic excision (TSME)? Participants will include patients who underwent curative right hemicolectomy for right-sided colon cancer between 2015 and 2020 at eight institutions. They will be categorized into two groups based on the surgical technique received-CME group and TSME group-and evaluated for primary and secondary endpoints of 5-year recurrence-free survival (RFS) and overall survival (OS), respectively.

DETAILED DESCRIPTION:
This observational, population-based cohort study was conducted following the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines, with approval obtained from the institutional review board (IRB) of the primary institution and the ethics committees of each participating institution in the Republic of Korea, Hong Kong, and Taiwan. Given that the study utilized anonymized retrospective data, the requirement for informed consent was waived.

The study aimed to evaluate the efficacy and safety of Tumor Specific Mesocolic Excision (TSME) compared to Complete Mesocolic Excision (CME) in patients with right-sided colon cancer. Patients diagnosed with right-sided colon cancer who underwent laparoscopic or robotic right hemicolectomy between 2015 and 2020 were included. Surgical techniques were classified into modified TSME or CME, and the study assessed oncologic outcomes, including recurrence-free survival (RFS), overall survival (OS), lymph node yield, and stage distribution.

Data collection was conducted at multiple medical centers across Asia to ensure a diverse representation of patient demographics and clinical practices. The participating institutions included Asan Medical Center, Korea University Anam Hospital, Severance Hospital, Kyungpook National University Chilgok Hospital, Chinese University of Hong Kong, North District Hospital, Pamela Youde Nethersole Eastern Hospital, and China Medical University Hospital. These centers, varying in location and size, enhance the study's generalizability within the context of right-sided colon cancer management in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic or robotic right hemicolectomy from 2015 to 2020
* Patients who received curative right hemicolectomy with lymphadenectomy

Exclusion Criteria:

* Familial adenomatous polyposis (FAP)
* Hereditary non-polyposis colon cancer (HNPCC)
* Patients with inflammatory bowel disease
* Patients with synchronous malignancies in other organs
* Patients with non-adenocarcinoma histology of colon cancer
* Patients with follow-up duration of less than 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included patients who underwent laparoscopic or robotic right hemicolectomy from 2015 to 2020 at 8 instituions : Asan Medical Center, Korea University Anam Hospital, Severance Hospital, Kyungpook National University Chilgok Hospital, Chinese University of Hong Kong, North District Hospital, Pamela Youde Nethersole Eastern Hospital, and China Medical University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3326 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
5 year Recurrence free survival | Outcome measures will be assessed at 5 years post-surgery.
  Recurrence-Free Survival (RFS) between patients who underwent TSME and CME procedures from 2015 to 2020

SECONDARY OUTCOMES:
Overall survival | Outcome measures will be assessed at 5 years post-surgery.
  Overall survival (OS) between patients who underwent TSME and CME procedures form 2015 to 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No